CLINICAL TRIAL: NCT00735384
Title: Application of Methodology of Non-invasive Stimulated Muscle Force Assessment to ICU Patients and Patients With Primary Myopathies to Characterize Their Muscle Weakness - Extension of the Study Protocol: 2008 to 2018
Brief Title: Muscle Force Assessment in the Intensive Care Unit and in Primary Myopathies
Status: Completed | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Collaborators: University of Minnesota (Other)
Responsible Party: Sponsor
Other Study IDs: 134/02; P21/08//A05/08 (Other: Else-Kröner-Fresenius-Stiftung 2008; SGAR / SSAR Fonds 2007, Schweizerische Muskelstiftung (SMS) 2016)
Record Dates: First submitted 2008-08-13; First posted 2008-08-14 (Estimated); Last update posted 2021-11-29 (Actual); Status verified 2021-11

CONDITIONS: Sepsis; Primary Myopathies
Keywords: sepsis; critical illness; muscle, skeletal; myopathy; isometric contraction; intensive care units; torque; muscular atrophy; malignant hyperthermia; skin resistance
MeSH Terms: conditions — Sepsis; Critical Illness; Muscular Diseases; Muscular Atrophy; Malignant Hyperthermia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Patients with critical illness myopathy: Patients with,e.g., sepsis, with secondary myopathy
- Patients with Primary Myopathies: Patients with primary myopathy, e.g., Duchenne Muscular Dystrophy, Myotonia

SUMMARY:
The primary aim of the project is to apply the non-invasive stimulated muscle force assessment system to i) intensive care unit patients and ii) patients with primary myopathy or subclinic myopathy (e.g., Duchenne muscular dystrophy, Myotonia, MH). The investigators will use this new methodology of force assessment to phenotype patients weakness during their illnesses (depict typical force pattern) and monitor recovery periods, or disease progression, respectively. This new system will be evaluated until the year 2018. The investigators will determine variables of isometric skeletal muscle force.

These systems should serve as force monitoring tools and help to guide therapies.

DETAILED DESCRIPTION:
A force measuring system similar to one employed in previous studies will be redesigned with a new stimulator system and leg support system. This new, small, light and portable measurement system accurately measures patients' muscle forces. The system produces repeatable results. Over a long-time time period, this system will be applied to ICU patients and patients with primary myopathies, e.g. muscular dystrophy Duchenne or myotonias, and their ankle dorsiflexor isometric torques measured after electrical peroneal nerve stimulation. Torques will be amplified and converted into electrical signals by a Whetstone bridge, and data will be stored on a computer (LabView system). Stimulated torque responses will be obtained regularly, and subsequently the individualized curves will be determined. Electromyogram will be performed at each recording session. For all subjects possible, the investigators will continue to monitor their stimulated muscle forces during their recovery periods or disease progression. Type of data: Variables of isometric skeletal muscle contractions, such as peak torques, contraction and relaxation times and torque latencies. To find an assumed difference of 50% in strength, at least 30 individuals (power 0.9) are required.

Values will be compared to patients voluntary forces, determined by Muscle Research Council (MRC) and Manual Muscle Test (MMT) scores.

Additionally, skin resistances of edema patients will by determined employing a twitch stimulator and an oscilloscope. We are interested whether edema (fluid) changes tissue resistance. Data are required to redesign the new stimulation unit of the muscle force measuring system.

ELIGIBILITY:
Inclusion Criteria:

* Any patient which fulfills the criteria for sepsis / septic shock according the definition of the American College of Chest Physicians/Society of Critical Care Medicine Consensus Conference
* Patients who will be sedated, mechanically ventilated, and immobilized
* Patients will be intubated the day of admission to ICU and started mechanically ventilated on a positive pressure ventilation modus
* The severity of each patient¢s illness will be assessed using the Acute Physiology and Chronic Health Evaluation (APACHE) II score with required entry scores of a minimum of 15-20 Points
* Patients suffering from a primary myopathy, e.g., Duchenne Muscular Dystrophy or subclinic myopathy, e.g. Malignant Hyperthermia.

Exclusion Criteria:

* Patients with neuropathies, consuming diseases in an advanced state (metastatic cancer) and severe infectious diseases (e.g. AIDS, Hepatitis), as well as patients with injured legs and/or patients requiring neuromuscular blocking drugs.
* Patients under the age of 18 yr.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Primary care clinic
Sampling Method: Non-Probability Sample
Enrollment: 22 (Actual)
Dates: Start 2006-09-01 (Actual); Primary Completion 2019-12-30 (Actual); Study Completion 2019-12-30 (Actual)

PRIMARY OUTCOMES:
Skeletal Muscle Force in ICU Patients and Patients with Primary Myopathies | ICU patients: 1-3 months; Myopathy patients: up to 5 years
  Characterisation and follow up of the muscle force of the lower leg in severly ill patients of a intensive-care-unit. To characterise primary myopathy patients typical force pattern of the lower leg and to follow up their individual disease progression over many years

SECONDARY OUTCOMES:
Muscle forces pending on the Malignant Hyperthermia (MH) status of a patient (susceptible to MH or not susceptible to MH) | at the time point of MH testing, i.e., at hospital admission

CONTACTS AND LOCATIONS:
Overall Officials: Albert Urwyler, Professor MD, Study Director — Departments of Anaesthesia and Research, University Hospital Basel
Locations (1):
- University of Basel Hospital, Basel, Switzerland

REFERENCES:
- [Result] Ginz HF, Iaizzo PA, Urwyler A, Pargger H. Use of non-invasive-stimulated muscle force assessment in long-term critically ill patients: a future standard in the intensive care unit? Acta Anaesthesiol Scand. 2008 Jan;52(1):20-7. doi: 10.1111/j.1399-6576.2007.01427.x. Epub 2007 Aug 20. PMID 17714574
- [Result] Ginz HF, Bandschapp O, Urwyler A, Girard T, Iaizzo PA. Tissue oedema is not associated with skeletal muscle weakness in septic patients. Acta Anaesthesiol Scand. 2010 Aug;54(7):904. doi: 10.1111/j.1399-6576.2010.02257.x. No abstract available. PMID 20649524
- [Result] Durfee WK, Young JR, Ginz HF. Inter-electrode tissue resistance is not affected by tissue oedema when electrically stimulating the lower limb of sepsis patients. J Med Eng Technol. 2014 May;38(4):227-31. doi: 10.3109/03091902.2014.904451. PMID 24758395
- [Result] Ginz HF, Iaizzo PA, Schweikert K, Durfee WK. Isometric skeletal muscle force measurement in primary myopathies. Muscle Nerve. 2016 Jun;53(6):913-7. doi: 10.1002/mus.24954. Epub 2016 Feb 8. PMID 26506402
- [Derived] Ginz HF, Iaizzo PA, Schweikert K, Durfee WK. Long-term monitoring of stimulated lower leg skeletal muscle forces compared with voluntary contractions in myopathy patients - A five-year follow-up report on 5 adults. J Bodyw Mov Ther. 2024 Apr;38:8-12. doi: 10.1016/j.jbmt.2024.01.011. Epub 2024 Jan 23. PMID 38763619